CLINICAL TRIAL: NCT04538404
Title: Score for the Prediction of Mortality Risk After Surgery for Colon Cancer in a Case Series of Elderly Patients
Brief Title: Mortality Score in Elderly Patients With Colon Cancer
Acronym: MECC
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Marialuisa Lugaresi, Adjunct Professor MD, PhD, University of Bologna
Other Study IDs: MECC Score
Record Dates: First submitted 2020-08-22; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Mortality; Surgery; Colon Cancer
Keywords: colon cancer; surgery; mortality; elderly; scoring system
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colon Surgery — Right, left colon surgery, transverse colon surgery, multiple colon surgery in open and minimally invasive surgert

SUMMARY:
CR-POSSUM is one of the most used surgical scores to predict mortality after colorectal surgery. Its main drawback is the requirement of intraoperative variables, whose collection is time-consuming and prevents from obtaining a purely preoperative risk assessment. The primary aim of the study is to develop a new surgical score using preoperative parameters to predict 30-day mortality after colon cancer surgery in the elderly population. The secondary objective is to analyze its efficacy compared to CR-POSSUM.

DETAILED DESCRIPTION:
Patients aged 80 and older undergoing surgery for colon cancer from 2011 to 2017 in an Italian hospital were retrospectively selected. MECC score [Mortality in Elderly patients with Colon Cancer] was calculated summing up the scores relating to: arterial saturation of O2, Systolic Blood Pressure, Heart Rate, WBCs, Albumin, Creatinine. Once CR-POSSUM was calculated, the two scores were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 80 and above having elective and emergency colonic resection for colon cancer via open, laparoscopic and converted approaches

Exclusion Criteria:

* Surgical resections for rectal cancer and surgical procedures for non-neoplastic colon pathologies

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Men and women patients aged 80 and above having elective and emergency colonic resection for colon cancer via open, laparoscopic and converted approaches.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
New surgical score using preoperative parameters to predict 30-day mortality after colon cancer surgery in the elderly population | Up to 30 days after surgery
  MEC Score (arterial saturation of O2, Systolic Blood Pressure, Heart Rate, WBCs, Albumin, Creatinine) for the evaluation of the risk of in-hospital mortality occurred during hospitalization up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Nardo, MD,PhD, Study Director — University of Bologna
Locations (2):
- Italy (2):
  - Bruno Nardo, Bologna
  - Marialuisa Lugaresi, Bologna

IPD SHARING:
Plan to Share IPD: No